CLINICAL TRIAL: NCT03784040
Title: da VINci Study (OTSGC-A24 Therapeutic Peptide Vaccine + Ipilimumab + Nivolumab) Nivolumab, Ipilimumab and OTSGC-A24 Therapeutic Peptide Vaccine in Gastric Cancer - a Combination Immunotherapy Phase Ib Study.
Brief Title: Nivolumab, Ipilimumab and OTSGC-A24 Therapeutic Peptide Vaccine in Gastric Cancer - a Combination Immunotherapy Phase Ib Study.
Acronym: da VINci
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: OncoTherapy Science, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA01/03/18; 2018/00422 (Other: NHG Domain Specifics Research Board)
Record Dates: First submitted 2018-12-20; First posted 2018-12-21 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer
Keywords: Nivolumab; Ipilimumab; OTSGC-A24
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Arm A) OTSGC-A24 + nivolumab (Experimental): Study subjects will receive nivolumab 240 mg intravenously (IV) and OTSGC-A24 consisted of 1 μmol (~1 mg) of OTSGC-A24-Fo, OTSGC-A24-De, OTSGC-A24-Ki, OTSGC-A24-VE1 and OTSGC-A24-Ur 1.0 μmol (as API) administered subcutaneously on Day 1 and D14 each 28 day cycle (q28d) for up to 24 months.
  Interventions: Drug: OTSGC-A24; Drug: Nivolumab
- (Arm B) OTSGC-A24 + nivolumab + ipilimumab (Experimental): Study subjects will receive nivolumab 240 mg intravenously (IV) and OTSGC-A24 consisted of 1 μmol (~1 mg) of OTSGC-A24-Fo, OTSGC-A24-De, OTSGC-A24-Ki, OTSGC-A24-VE1 and OTSGC-A24-Ur 1.0 μmol (as API) administered subcutaneously on Day 1 and D14. Ipilimumab 1mg/kg (IV) will be administered q6w (i.e. C1D1, C2D15, C3D1 …) of each 28 day cycle for up to 24 months.
  Interventions: Drug: OTSGC-A24; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: OTSGC-A24 — OTSGC-A24 is administered as a subcutaneous (under the skin) injection. Nivolumab and ipilimumab are administered by intravenous (IV) infusion, meaning the drug is given through a catheter in a vein. A pump will be used to ensure the correct amount of medicine is given through the catheter. The nivolumab and ipilimumab infusions each take about 30 minutes. There will be a break of about 30 minutes in between the nivolumab and ipilimumab infusions (if given on the same day). OTSGC-A24 and nivolumab are administered every 2 weeks, while ipilimumab is administered every 6 weeks.
Drug: Nivolumab — OTSGC-A24 is administered as a subcutaneous (under the skin) injection. Nivolumab and ipilimumab are administered by intravenous (IV) infusion, meaning the drug is given through a catheter in a vein. A pump will be used to ensure the correct amount of medicine is given through the catheter. The nivolumab and ipilimumab infusions each take about 30 minutes. There will be a break of about 30 minutes in between the nivolumab and ipilimumab infusions (if given on the same day). OTSGC-A24 and nivolumab are administered every 2 weeks, while ipilimumab is administered every 6 weeks.
Drug: Ipilimumab — OTSGC-A24 is administered as a subcutaneous (under the skin) injection. Nivolumab and ipilimumab are administered by intravenous (IV) infusion, meaning the drug is given through a catheter in a vein. A pump will be used to ensure the correct amount of medicine is given through the catheter. The nivolumab and ipilimumab infusions each take about 30 minutes. There will be a break of about 30 minutes in between the nivolumab and ipilimumab infusions (if given on the same day). OTSGC-A24 and nivolumab are administered every 2 weeks, while ipilimumab is administered every 6 weeks.
  Arms: (Arm B) OTSGC-A24 + nivolumab + ipilimumab

SUMMARY:
The primary hypothesis is that cancer vaccine can convert non-immunogenic gastric cancer into immunogenic phenotype susceptible to PD1 inhibition. This would lead to an improved radiological response rate and favorable immune contexture for immune checkpoint blockade

DETAILED DESCRIPTION:
Primary Objectives

1. Safety cohorts: To evaluate the safety of OTSGC-A24 and nivolumab (+ ipilimumab) in patients with refractory gastric cancer.
2. Arm A: To determine the objective response rate of OTSGC-A24 and nivolumab in advanced gastric cancer.
3. Arm B: To determine the objective response rate of OTSGC-A24 and nivolumab + ipilimumab in advanced gastric cancer.

Secondary Objectives

1. To compare the difference in objective response rates between Arm A and Arm B
2. To compare the tumoral immune contexture and PDL-1 expression before treatment, after OTSGC-A24, and after nivolumab (+ ipilimumab) in combination with OTSGC-A24.
3. To determine the serum cytotoxic T-cell response using enzyme-linked immunospot assay (ELISPOT) in PBMC.
4. To determine the progression-free survival (PFS) and overall survival (OS) of Arm A and Arm B.
5. To evaluate the effect of OTSGC-A24 and nivolumab + ipilimumab on clinical and immune PD markers.
6. Evaluate the effects of treatment on peripheral T-cell phenotypic profiles with epitope-specificities by coupling mass cytometric analyses with highly-multiplexed peptide-MHC tetramer staining technology.
7. Identify potential biomarkers for treatment response and mechanisms of secondary resistance by studying gene expression profiles and phenotypic/functional markers of tumour and infiltrating immune cells.

End Points - Efficacy

The endpoints for efficacy are:

* Induction of specific CTL response after vaccination
* Response rate
* Progression-free survival
* Overall survival End Points - Safety

The endpoints for safety are:

• overall adverse events observed, treatment-related adverse events, and category (eg percentage of patients with any-grade treatment-related adverse events and grade 3-4 treatment-related adverse events).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed inoperable or metastatic gastric cancer that has failed or demonstrated intolerance to standard therapy - which includes platinum or fluoropyrimidine or taxane based chemotherapy.
2. Patients must have measurable disease.
3. Age ≥ 21 years
4. ECOG performance status (PS) of 0 to 1
5. Life expectancy at least 3 months
6. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) ≥ 1,500/mcL
   * Platelets ≥ 100,000/mcL
   * Total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
   * Creatinine <1.5x normal institutional limits
7. Patients must be HLA-A*24:02
8. Patients must have recovered (< grade 1) from all reversible treatment toxicity from prior chemotherapy, radiotherapy or surgery.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients receiving any other investigational products
2. Patients who have previously received prior nivolumab or PD-/L1 blockade therapy
3. Active autoimmune disease requiring disease-modifying therapy.
4. Concurrent systemic steroid therapy higher than physiologic dose (equivalent of prednisolone 10mg daily)
5. Any form of active primary or secondary immunodeficiency.
6. History of significant gastrointestinal bleeding that required intervention within the prior 1 month is ineligible; inherited bleeding diathesis or coagulopathy.
7. Serious non healing wound and peptic ulcer disease
8. Previous history of intestinal perforation
9. Symptomatic central nervous system (CNS) metastasis
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension (systolic >160 mmHg and/or diastolic >100 mmHg), symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction/cerebrovascular event (≤ 6 months prior to study entry), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, long term systemic immunosuppressant or corticosteroid, and active viral hepatitis.
11. Women who are breast-feeding or pregnant are excluded from this study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event and Adverse Drug Reaction | 3 years
Response Rate | 3 years

SECONDARY OUTCOMES:
Rate of induction of specific CTL response | 3 years
Progression-free Survival | 3 years
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Background] Janunger KG, Hafstrom L, Nygren P, Glimelius B; SBU-group. Swedish Council of Technology Assessment in Health Care. A systematic overview of chemotherapy effects in gastric cancer. Acta Oncol. 2001;40(2-3):309-26. doi: 10.1080/02841860151116385. PMID 11441938